CLINICAL TRIAL: NCT06041191
Title: An Investigation of Sensory Processing Skills in Toddler With Joint Hypermobility
Brief Title: Sensory Processing Skills in Toddler With Joint Hypermobility
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayse Simsek, assistant professor, Gazi University
Other Study IDs: E-77082166-604.01.02-687785
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Child Development; Sensory Disorder; Hypermobility, Joint
MeSH Terms: conditions — Sensation Disorders; Joint Instability | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with GJH: Children who scored above 4 points in the hypermobility assessment made with the Beighton score were included in this group. sensory processing skills assessed with the Test of Sensory Functions in Infants
  Interventions: Diagnostic Test: Assessment
- Children without GJH: Children who scored below 4 points in the hypermobility assessment made with the Beighton score were included in this group. sensory processing skills assessed with the Test of Sensory Functions in Infants
  Interventions: Diagnostic Test: Assessment

INTERVENTIONS:
Diagnostic Test: Assessment — The children included in the study were evaluated in terms of hypermobility and then divided into two groups. Children in both groups were evaluated in terms of sensory processing skills.

SUMMARY:
shows that children and adults with joint hypermobility may be identified with common clinical problems that are unrelated, such as chronic fatigue, anxiety, and a range of gastrointestinal functional disorders [4-6]. Considering the relationship of joint hypermobility with joint muscle tone and posture, sensory processing skills may also be affected in individuals with hypermobility. No study in the literature examines the relationship between joint hypermobility and sensory processing. This study was planned to detect joint hypermobility as early as 12-14 months and to examine its relationship with sensory processing skills.

ELIGIBILITY:
Inclusion Criteria:

12-14 month old healthy children

-

Exclusion Criteria:

* they had major congenital malformations, had genetic or chromosomal abnormalities, had known metabolic disorders, or had seizures.

Ages: 12 Months to 14 Months | Sex: All
Age Groups: Child
Study Population: Healthy children born at term between 12-14 months
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Beighton Score | 20minutes
  . The test consists of 5 items: (1) positive if the passive dorsiflexion of the fifth metacarpophalangeal joint score is greater than 90 degrees (bilateral test); (2) positive if passive hyperextension of the elbow joint is >10 (bilateral test); (3) positive if passive hyperextension of the knee joint is >10 (bilateral test); (4) passive apposition of the thumb to the flexor side of the forearm is positive for joint hypermobility (bilateral test) if the shoulder is at 90 flexion, the elbow is extended, and the whole thumb is touching the flexor side of the forearm; and (5) the score is positive when dorsiflexion of the ankle is >30 (bilateral test). The assessment was performed on both the right and left sides, and the item was given 1 point if hypermobility was detected in the joints, and 0 points if not, according to the instructions of each item. Cut-off score of >4 was used to define hypermobility

SECONDARY OUTCOMES:
Test of Sensory Functions in Infants | 20 minutes
  The TSFI is primarily used to assess sensory defense behaviors in infants aged 4-18 months. Test; It consists of 5 subsections and 24 items. TSFI requires the infant to be stimulated and interact with a variety of materials. The total score varies between 0-49 and the test has norm values for different age groups. Although it is used from the fourth month, the most reliable and valid results are obtained between 7-18 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University, Erzurum, Turkey (Türkiye)